CLINICAL TRIAL: NCT06860282
Title: A Phase I, Randomized, Parallel-Controlled, Single and Multiple Ascending Dose Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of CX2101A Enteric-Coated Tablets in Healthy Chinese Adult Subjects
Brief Title: A Study of CX2101A Enteric-Coated Tablets in Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heronova Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHRC-CX2101-01
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Coronavirus Pneumonia
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Masking Description: Part 1 is open label, Part 2 is double-blinded (participant and investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- SAD,Remdesivir (Active Comparator): Participants received single dose of intravenous remdesivir.
  Interventions: Drug: Remdesivir
- SAD,CX2101A (Experimental): Participants received single dose of CX2101A orally. Dose levels are 20 mg, 80 mg, 160 mg, 300 mg and 600 mg.
  Interventions: Drug: CX2101A
- MAD,Placebo (Placebo Comparator): Participant received CX2101A placebo matching CX2101A orally once daily for 5 days.
  Interventions: Drug: Placebo
- MAD, CX2101A (Experimental): Participant received CX2101A orally once daily for 5 days. Dose levels are 100 mg and 300 mg.
  Interventions: Drug: CX2101A
- FE, CX2101A (Experimental): Participants received single dose of CX2101A 300 mg orally under fed conditions.
  Interventions: Drug: CX2101A

INTERVENTIONS:
Drug: Remdesivir — Intravenous remdesivir 100 mg
  Arms: SAD,Remdesivir
Drug: CX2101A — CX2101A enteric-coated tablet
  Arms: FE, CX2101A; MAD, CX2101A; SAD,CX2101A
Drug: Placebo — CX2101A placebo enteric-coated tablet
  Arms: MAD,Placebo

SUMMARY:
This study is divided into two parts, including Part I: a randomized, open-label, positive drug-controlled, single ascending dose (SAD) study, a food effect (FE) study, and Part II: a randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study.

DETAILED DESCRIPTION:
Part I: Single Ascending Dose (SAD) and Food Effect (FE) Study Combined SAD and FE Study (N=42): The SAD portion is integrated with the FE study, comprising 5 dose groups: 20 mg, 80 mg, 160 mg, 300 mg, and 600 mg. The trial commences with the low-dose group and in a sequential manner. As subjects in a given dose group of CX2101A complete their safety assessments, the investigator evaluates whether the low-dose group has met the dose-escalation termination criteria. If not, the trial escalates to the next dose level.

SAD Study Enrollment: The SAD study aims to enrolls a total of 42 healthy subjects. The 20 mg dose group will enroll 4 subjects, while the 80 mg, 160 mg, and 600 mg dose groups will each enroll 8 subjects. These subjects will be randomly assigned to receive either CX2101A enteric-coated tablets or intravenous remdesivir in a 3:1 ratio.

FE Study for the 300 mg Dose Group: The 300 mg dose group will concurrently conduct a study of food effect on the pharmacokinetics (PK) of CX2101A enteric-coated tablets. This study plans to enroll 14 subjects, who will be randomly assigned to receive either CX2101A enteric-coated tablets (12 subjects) or intravenous remdesivir (2 subjects). In the first period, all 14 subjects will receive a single dose under fasting conditions according to the randomization schedule and will have blood samples collected. The 12 subjects receiving CX2101A enteric-coated tablets will undergo a 7-day washout period with a potential adjustment based on PK data from prior dose groups before proceeding to the second period, where they will receive the drug under fed conditions, complete blood sample collection, and undergo safety assessments.

Part II: Multiple Ascending Dose (MAD) Study MAD Study Design: The MAD study will include 2 dose groups, 100 mg and 300 mg. It plans to enroll 20 healthy adult subjects, with 10 subjects in each dose group. These subjects will be randomly assigned to receive either CX2101A enteric-coated tablets (8 subjects) or CX2101A placebo (2 subjects). The study will involve continuous dosing for 5 days. If the subjects in the first dose group complete their safety assessments and the investigator determines that the dose-escalation termination criteria have not been met, the study will escalate to the next dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between 18 and 55 years old (including 18 and 55 years old), regardless of gender.
2. For male volunteers, the body weight should be ≥ 50.0 kg, and for female volunteers, the body weight should be ≥ 45.0 kg. The body mass index (BMI) = body weight (kg) / height² (m²), and it should be within the range of 19.0 to 28.0 kg/m². Women of childbearing potential (WOCBP) or the female partners of male subjects should be willing to have no plans for childbearing from 2 weeks before the screening until 3 months after the last administration of the investigational medicinal product, and voluntarily adopt effective contraceptive measures (including one or more non-pharmacological contraceptive measures), and have no plans for sperm donation or egg donation.
3. No history of major diseases, and the results of physical examination, vital signs, 12-lead electrocardiogram, chest X-ray examination and laboratory tests during the screening period are normal, or although slightly beyond the normal reference value range, they are judged by the investigator to have no clinical significance.
4. The subject should be able to maintain good communication with the investigator, comply with various requirements of the clinical trial, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Diseases with abnormal clinical manifestations that occurred before screening or are currently occurring and need to be excluded, including but not limited to those in the nervous/mental system, respiratory system, cardiovascular and cerebrovascular system, digestive system (any history of gastrointestinal diseases that affect drug absorption), hematological and lymphatic system, urinary system, endocrine system, and immune system.
2. Acute diseases that occurred from the screening stage to before the administration of the investigational medicinal product and are judged by the investigator to possibly affect the research results.
3. Subjects who cannot tolerate intravenous puncture or those with a history of syncope judged by the investigator to be of clinical significance.
4. Subjects with difficulty in swallowing.
5. Subjects who are judged by the investigator to possibly or definitely have an allergic reaction to the investigational drug, remdesivir (including similar drugs), or any of its excipients; or subjects with an allergic constitution judged by the investigator to be of clinical significance (a history of severe allergies to multiple drugs and foods) or a history of allergic diseases.
6. Subjects who have undergone surgery before screening and are judged by the investigator to possibly affect the absorption, distribution, metabolism, and excretion of the drug, or subjects with severe surgical sequelae, or subjects who plan to undergo surgery during the study period.
7. Subjects who donated blood or had massive blood loss (≥ 400 mL), donated ≥ 2 units of component blood, or received a blood transfusion within 3 months before the first administration of the trial, or those who plan to donate blood during the trial.
8. Subjects who received any investigational drug in a clinical study or participated in any interventional clinical study within 3 months before the first administration of the trial.
9. Subjects who smoked an average of more than 5 cigarettes per day within 3 months before the first administration of the trial, or those who cannot stop using any tobacco products during the trial.
10. Subjects who consumed an average of more than 14 units of alcohol per week within 3 months before the first administration of the trial (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with an alcohol content of 40% or 150 mL of wine), or those who cannot stop using any alcohol-containing products during the trial, or those with a positive alcohol breath test before the administration of the trial.
11. Subjects who consumed an excessive amount of tea, coffee, and/or caffeine-containing beverages on average per day (more than 8 cups on average, 1 cup ≈ 250 mL) within 3 months before the first administration of the trial, or those who cannot stop consuming tea, coffee, and/or caffeine-containing beverages during the trial.
12. Subjects who used any prescription drugs, over-the-counter drugs, traditional Chinese patent medicines, Chinese herbal medicines, vitamins, or health foods within 28 days before screening or within 5 drug half-lives (whichever is longer).
13. Female subjects who are pregnant or breastfeeding, or those with a positive blood/urine pregnancy test (only for WOCBP) at any time before the first administration.
14. Positive results or results exceeding the upper limit of the reference range for the four hemodialysis tests: hepatitis B surface antigen (HBsAg), quantitative hepatitis C (HCV) antibody, quantitative human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody.
15. Subjects with a positive urine drug screening (morphine, tetrahydrocannabinolic acid, methamphetamine, methylenedioxymethamphetamine, ketamine) or those with a history of drug abuse or drug use within the past 5 years before the trial.
16. Subjects who consumed or drank pitaya, mango, pomelo, carambola, or foods or beverages prepared from them, or foods or beverages containing xanthine, caffeine, or alcohol (including chocolate, tea, coffee, cola, cocoa, etc.), or other special diets that affect the absorption, distribution, metabolism, and excretion of the drug within 72 hours before the first administration.
17. Subjects with special dietary requirements, lactose intolerance, or those who cannot accept the unified diet.
18. Subjects who, according to the investigator's judgment, are not suitable to participate in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Rate and severity of treatment-emergent adverse events (TEAEs) | From day 1 until 5 days after treatment
  Based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Vital signs | From day 1 until 5 days after treatment
  Assessment of blood pressure
Vital signs | From day 1 until 5 days after treatment
  Assessment of heart rate
Vital signs | From day 1 until 5 days after treatment
  Assessment of respiratory rate
Vital signs | From day 1 until 5 days after treatment
  Assessment of body temperature.
Electrocardiogram (ECG) | From day 1 until 5 days after treatment
  ECG QT Interval
Physical examinations | From day 1 until 5 days after treatment
  Assessment of head, eyes, ears, nose, and throat, chest, cardiac, abdominal, extremities, neurologic, and lymph node examinations
Complete blood count test | From day 1 until 5 days after treatment
  Assessment includes Platelet Count, Hemoglobin, WBC Count (absolute), Neutrophils, Lymphocytes, Eosinophils, Monocytes, Basophils
Clinical Chemistry | From day 1 until 5 days after treatment
  Assessment includes BUN, Creatinine, Glucose (fasting), Sodium, Total Protein, Magnesium , Potassium, Chloride, Total CO2, Calcium, Albumin, AST (SGOT), ALT (SGPT), Phosphorous, Alkaline phosphatase, Total and direct bilirubin

SECONDARY OUTCOMES:
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Peak Concentration (Cmax): The maximum plasma concentration of the drug.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-t): The area under the plasma concentration-time curve from time zero to the last measurable concentration.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Area Under the Curve from Time Zero Extrapolated to Infinity (AUC0-∞): The area under the plasma concentration-time curve from time zero extrapolated to infinity.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Time to Reach Peak Concentration (Tmax): The time at which the peak plasma concentration is reached.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Elimination Half-Life (T1/2): The time required for the plasma concentration to decrease by half.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Apparent Volume of Distribution (Vz/F): The volume into which the drug appears to be distributed, corrected for bioavailability.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Apparent Clearance (CL/F): The clearance of the drug from the plasma, corrected for bioavailability.
PK profile of CX2101A and its metabolite CX210101,CX210108, CX210144, remdesivir and its metabolite GS-441524 | From time zero up to 120 hours post-dose
  Percentage of AUC Extrapolated (AUC_%Extrap): The percentage of the total AUC that is extrapolated beyond the last measurable concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No